CLINICAL TRIAL: NCT02965443
Title: Effectiveness of Dapagliflozin + Saxagliptin to Revert From a Basal-bolus Insulin Treatment (BBIT) Regimen to a Basal Supported Oral Therapy (BOT) in Patients With Type 2 Diabetes
Brief Title: Dapagliflozin + Saxagliptin in a Basal-bolus Insulin Treatment
Acronym: DapaSaxaBBIT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low patient recruitment
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UTUB - 2015-005740-34
Record Dates: First submitted 2016-10-28; First posted 2016-11-16 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2018-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Active Comparator): Dapagliflozin 10 mg + Saxagliptin 5 mg, each once daily, for 24 weeks
  Interventions: Drug: Dapagliflozin 10 mg + Saxagliptin 5 mg
- Placebo (Placebo Comparator): Placebo 1 10 mg + Placebo 2 5 mg, each once daily, for 24 weeks
  Interventions: Drug: Placebo 1 10 mg + Placebo 2 5 mg

INTERVENTIONS:
Drug: Dapagliflozin 10 mg + Saxagliptin 5 mg — 24 weeks intervention with Dapagliflozin 10 mg + Saxagliptin 5 mg
  Other Names: Forxiga + Onglyza
  Arms: Verum
Drug: Placebo 1 10 mg + Placebo 2 5 mg — 24 weeks intervention with Placebo 1 10 mg + Placebo 2 5 mg
  Other Names: Placebo 1 + Placebo 2
  Arms: Placebo

SUMMARY:
To perform a study that investigates the effectiveness of adding the SGLT2 inhibitor dapagliflozin + the dipeptidyl peptidase 4 (DPP-4) inhibitor saxagliptin vs placebo to revert from a BBIT regimen to a BOT regimen in patients with type 2 diabetes.

DETAILED DESCRIPTION:
This will be a phase IV study investigating the efficacy and safety of adding the SGLT2 inhibitor dapagliflozin together wih the DPP-4 inhibitor saxagliptin to an intensified insulin treatment regimen. Because BOT is superior to BBIT in respect to the development of bodyweight, hypoglycaemia and patient satisfaction in type 2 diabetes, we hypothesize that the combined addition of the SGLT2 inhibitor dapagliflozin with the DPP-4 inhibitor saxagliptin is effective and safe to revert from a BBIT to a BOT treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Age 18 - 75 years
* Anti-GAD antibodies negative (Glutamic Acid Decarboxylase)
* C-peptide levels ≥ 1.5 ng/mL
* Fasting blood glucose > 126 mg/dl
* HbA1c 8.0 - 10.5 %
* BMI 25.0 - 45.0 kg/m2
* Previous therapy with BBIT (basal insulin and at least once daily bolus insulin)

Exclusion Criteria:

* Use of any oral antidiabetic treatment except for metformin (i.e., sulphonylureas, DPP-IV inhibitors, thiazolidinediones, SGLT-2 inhibitors (Sodium dependent glucose transporter) or GLP-1 analogues (glucagone like peptide) within the last three months prior to Screening
* Repeated episodes of severe hypoglycaemia within the last six months prior to Screening
* History of diabetic ketoacidosis, precoma diabetica, or diabetic coma
* Treatment with any other investigational drug within the last three months before Screening
* Acute infections within the last four weeks prior to Screening
* Recurrent urogenital infections
* History of pancreatitis
* Anamnestic history of hypersensitivity to the study drugs or to drugs with similar chemical structures
* History of severe or multiple allergies
* Concomitant participation in other clinical trials
* Type 1 diabetes
* Cardiovascular disease Clinically relevant ventricular tachycardia or ventricular fibrillation, 3rd degree AV block or Torsades de Pointes or treatment with antiarrhythmic drugs. Percutaneous coronary intervention within the past 6 months. Any of the following within the past 6 months: myocardial infarction (MI), coronary artery bypass surgery; unstable angina; or stroke.

Uncontrolled unstable angina pectoris or history of pericarditis, myocarditis, endocarditis. Congestive heart failure NYHA (New York Heart Association) class III or IV. Increased risk of thromboembolism, e.g. subjects with a history of deep leg vein thrombosis or family history of deep leg vein thrombosis, as judged by the Investigator.

* Malignancy including leukemia and lymphoma within the last 5y.
* Liver disease such as cirrhosis or chronic active hepatitis.
* Significant renal dysfunction (see also exclusion criteria laboratory abnormalities).
* State after kidney transplantation
* Endocrine disease:

Acromegaly or treatment with growth hormone or similar drugs. Chronic oral or parenteral corticosteroid treatment (>7 consecutive days of treatment) within 8 weeks; thyroid hormone replacement is allowed if the dosage has been stable for at least 3 months and the TSH is within normal limits

•Any of the following significant laboratory abnormalities: eGFR (as calculated by the MDRD equation) < 60 ml/min at Screening Fasting triglycerides >700 mg/dl (>7.9 mmol/l)

* Systolic blood pressure outside the range of 100-160 mmHg or diastolic blood pressure above 95 mmHg at Screening
* History of active substance abuse (including alcohol > 40g/day) within the past 2 years.
* Pregnancy or childbearing potential without adequate contraception
* Present therapy with systemic steroids
* Presence of psychiatric disorder or intake of anti-depressive or anti-psychotic agents with the exception of benzodiazepines and SSRIs/SNRI´s (selective serotonin reuptake inhibitor)
* Potentially unreliable subjects, and those judged by the investigator to be unsuitable for the study.
* Contraindications for Magnetic resonance (MR) scanning such as persons with cardiac pacemaker and implants out of metal or claustrophobia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving a HbA1c ≤ 7.5% and having a reversal from a BBIT to a BOT regimen | 24 weeks
  Percentage of subjects achieving a HbA1c ≤ 7.5% and having a reversal from a BBIT to a BOT regimen with treatment of dapagliflozin/saxagliptin or placebo

SECONDARY OUTCOMES:
changes in HbA1c between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in hypoglycaemic events between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in fasting blood glucose between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in daily insulin dose between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in bodyweight between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in body fat content between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in body fat distribution between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in liver fat content between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in intra-nasal insulin-induced brain fMR (functional magnetic resonance) imaging results between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in blood pressure between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in the blood lipid profile between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in microalbuminuria between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in well being and disease perception between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in fear of hypoglycemia between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo

OTHER OUTCOMES:
changes in fetuin-A levels between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in adiponectin levels between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in (Interleucin 1?ßß) IL-1ß levels between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in Il-6 levels between groups | 24 weeks
  treatment of dapagliflozin/saxagliptinn or placebo
differences in adverse events between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
differences in severe adverse events between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
differences in heart rate between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
differences in ECG parameters between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo
changes in clinical chemistry/haematology parameters between groups | 24 weeks
  treatment of dapagliflozin/saxagliptin or placebo

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No